CLINICAL TRIAL: NCT00166816
Title: The Pharmacokinetics and Dosage Regimen of Sirolimus in a Cyclosporine or Tacrolimus-Based Immunosuppression in Renal Transplant Patients
Brief Title: The Pharmacokinetics of Sirolimus When Combined With Cyclosporine or Tacrolimus in Renal Transplant Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 900604; NTUH S010
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2001-07

CONDITIONS: Transplantation; Kidney Transplantation; Immunosuppression
Keywords: Sirolimus; Tacrolimus; Cyclosporine; Pharmacokinetics; Immunosuppressive Agents; Immunosuppression; Kidney Transplantation; Transplantation
MeSH Terms: interventions — Sirolimus; Cyclosporine; Tacrolimus

INTERVENTIONS:
Drug: sirolimus, cyclosporine, tacrolimus

SUMMARY:
The purpose of this study is to understand the pharmacokinetic of sirolimus in different regimens, as well as the dose-level relationship of cyclosporine and tacrolimus, and design the most appropriate cyclosporine/sirolimus/steroid or tacrolimus/sirolimus/steroid dose regimen for Taiwanese.

DETAILED DESCRIPTION:
The dose and pharmacokinetic of an immunosuppressant may differ in different ethnics, and different combinations.

The purpose of this study is to determine the dose-level relationship of sirolimus through pharmacokinetic study. The dose-level relationship of cyclosporine and tacrolimus was also assessed. From clinical outcome and blood level of sirolimus and cyclosporine or tacrolimus, we can design the most appropriate cyclosporine/sirolimus/steroid or tacrolimus/sirolimus/steroid dose regimen for Taiwanese.

ELIGIBILITY:
Inclusion Criteria:

* De novo kidney transplantation patients, aged 13-65 years,have aminotransferase concentrations within 2 times the upper limit of normal.

Exclusion Criteria:

* pregnancy, tuberculosis, hepatitis B or C carrier status, human immunodeficiency virus-positive status, retransplantation or multiorgan transplantation, or history of rheumatoid arthritis.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2002-03; Study Completion 2003-06

PRIMARY OUTCOMES:
Pharmacokinetics of sirolimus in different regimens
Dose-concentration relationship of sirolimus

SECONDARY OUTCOMES:
Efficacy of rejection prevention
Dosage regimen of sirolimus + cyclosporine or tacrolimus
Dose-concentration relationship of cyclosporine/tacrolimus

CONTACTS AND LOCATIONS:
Overall Officials: Po-Huang Lee, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Wu FL, Tsai MK, Chen RR, Sun SW, Huang JD, Hu RH, Chen KH, Lee PH. Effects of calcineurin inhibitors on sirolimus pharmacokinetics during staggered administration in renal transplant recipients. Pharmacotherapy. 2005 May;25(5):646-53. doi: 10.1592/phco.25.5.646.63593. PMID 15899725
- [Derived] Tsai MK, Wu FL, Lai IR, Lee CY, Hu RH, Lee PH. Decreased acute rejection and improved renal allograft survival using sirolimus and low-dose calcineurin inhibitors without induction therapy. Int J Artif Organs. 2009 Jun;32(6):371-80. doi: 10.1177/039139880903200608. PMID 19670189